CLINICAL TRIAL: NCT07304921
Title: The Intake of Omega-3 Fatty Acids and the Inhibition of Their Mitochondrial Metabolism Increase EPA and DHA Levels in Healthy Volunteers
Brief Title: Novel Approach to Increase EPA and DHA Levels
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Riga Stradins University (Other)
Responsible Party: Principal Investigator, Ilze Konrade, PhD, MD, Riga Stradins University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: VPP-2022/1-000-28/2022
Record Dates: First submitted 2025-11-20; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Lipid Metabolism; Omega-3 Polyunsaturated Fatty Acids; Supplementation
Keywords: PUFA; meldonium; EPA; DHA; cardiometabolic health; acylcarnitines
MeSH Terms: interventions — 3-(2,2,2-trimethylhydrazine)propionate; Fatty Acids, Unsaturated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1: PUFAs supplementation only (Experimental): Participants received only PUFA supplements, metabolic parameters measured in plasma in the beginning, middle and end of study period
  Interventions: Dietary Supplement: PUFA supplementation only
- Arm 2: PUFAs followed by PUFAs+ meldonium (Experimental): Participants received PUFA supplements at the beginning, but after one month meldonium therapy was added to PUFA supplementation. Metabolic parameters measured in plasma in the beginning, middle and end of study period
  Interventions: Dietary Supplement: PUFA + meldonium
- Arm 3: Meldonium followed by meldonium+ PUFAs (Experimental): Participants received meldonium therapy at the beginning, but after one month PUFAs supplementation was added to meldonium therapy. Metabolic parameters measured in plasma in the beginning, middle and end of study period
  Interventions: Drug: Meldonium + PUFA

INTERVENTIONS:
Drug: Meldonium + PUFA — Meldonium (1g/day) or four weeks, followed by an additional four weeks of combined meldonium and PUFA (930 mg EPA and 750 mg DHA) supplement
  Arms: Arm 3: Meldonium followed by meldonium+ PUFAs
Dietary Supplement: PUFA + meldonium — PUFA supplement (930 mg EPA and 750 mg DHA) for four weeks, followed by an additional four weeks of combined PUFA supplement with 1 g/day meldonium
  Arms: Arm 2: PUFAs followed by PUFAs+ meldonium
Dietary Supplement: PUFA supplementation only — PUFA supplement containing 930 mg EPA and 750 mg DHA for 8 weeks
  Arms: Arm 1: PUFAs supplementation only

SUMMARY:
The goal of this intervention trial is to evaluate whether combining meldonium therapy with PUFAs (polyunsaturated fatty acids) supplements containing eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) changes the plasma (blood component) concentration of EPA and DHA, as well as the acylcarnitine (fatty acid metabolite) profile in healthy volunteers. The main questions it aims to answer are:

Does using meldonium together with PUFA supplements increase PUFA (EPA and DHA) concentrations in blood plasma? Does meldonium therapy change change the fatty acid metabolite (acylcarnitine) profile, if used together with PUFA supplements?

Researchers compared plasma metabolic parameters in the beginning, middle and end of study period in a group who received only PUFA supplements, with a group which got PUFA supplements at the beginning, but after one month meldonium therapy was added and a group which got meldonium therapy at the beginning, but after one month PUFA supplements were added.

Participants:

1. Received detailed information about the study and signed an informed consent form.
2. They were assigned to one of three study groups and received PUFAs and/or meldonium for the duration of the study.
3. Plasma samples were collected at the beginning, middle and end of the study period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults (age 18 and older)

Exclusion Criteria:

* Previously diagnosed serious chronic diseases (diabetes mellitus, atherosclerotic cardiovascular diseases, chronic kidney and liver diseases, cancer)
* PUFA supplement usage and/or meldonium therapy at least 6 months before inclusion in the study
* Participation in other clinical drug trials
* Pregnancy and breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-04-06 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Changes in the plasma concentrations of EPA and DPA | From enrollment moment to the end of 8 week study period
Changes in plasma acetylcarnitine concentrations | From the enrollment moment to the end of 8 week study period
  Acetylcarnitine contains acyl group with 2 carbon atoms
Changes in plasma medium-chain acylcarnitine concentration | From enrollment moment to the end of 8 week study period
  Medium- chain acylcarnitines are defined as containing acyl groups with 6-12 carbon atoms
Changes in plasma long-chain acylcarnitine concentration | Time Frame: From the enrollment moment to the end of 8 week study period
  Long-chain acylcarnitines contain acyl groups with 14-18 carbon atoms

SECONDARY OUTCOMES:
Changes in plasma meldonium concentration | From the enrollment moment to the end of 8 week study period
Changes in plasma gamma-butyrobetaine (GBB) concentrations | From the enrollment moment to the end of 8 week study period

CONTACTS AND LOCATIONS:
Overall Officials: Ilze Konrade, PhD, MD, Principal Investigator — Riga Stradins University
Locations (1):
- Riga Stradins university, Riga, Latvia

IPD SHARING:
Plan to Share IPD: Yes
We will deposit individual original measurement results, but not anthropometric data.
Supporting Information: Study Protocol
Time Frame: Available immediately following completion of the study. Study data will be stored indefinitely in accordance with institutional and regulatory requirements
Access Criteria: Data will be provided to researchers on request. We will evaluate whether their purpose comply with the consent and ethics approval.
URL: https://zenodo.org/records/16900133

REFERENCES:
- Available data/document: Individual Participant Data Set — https://zenodo.org/records/16900133